CLINICAL TRIAL: NCT03909113
Title: Tolerability of the New Hypoallergenic Formula in Children With IgE Mediated Cow's Milk Allergy
Brief Title: Tolerability of Hypoallergenic Formula in Children With Cow's Milk Allergy
Acronym: SINEALLII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Associate Professor, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 440/19
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Allergy Milk
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amino acid based formula (Experimental): amino acid based formula
  Interventions: Dietary Supplement: amino acid based formula

INTERVENTIONS:
Dietary Supplement: amino acid based formula — amino acid based formula

SUMMARY:
Cow's milk protein allergy is defined as an immunological reaction to one or more milk proteins. A variety of symptoms can be suggestive for cow's milk protein allergy . Cow's milk protein allergy is suspected clinically in 5-15% of infants, while most estimates of prevalence of cow's milk protein allergy vary from only 2 to 5 %. Confusion regarding cow's milk protein allergy prevalence is often due to differences in study populations, study design and a lack of defined diagnostic criteria. The importance of defined diagnostic criteria needs to be emphasised. It precludes infants from an unnecessary diet and avoids delay in diagnosis, which can lead to malnutrition. The treatment of cow's milk protein allergy is the dietary elimination of cow's milk proteins. In non-breastfed infants and children less than 2 years of age, a substitute formula is mandatory as prescribed by several international scientific societies. Extensively hydrolyzed formulas are used as therapeutic formulas. An extensively hydrolysed formula is often a whey or casein based formula in which the protein has been chopped up in smaller pieces that are less allergenic. Because of high cross-reactivity (up to 80%) and nutritional inadequacy, the use of any other animal milk or soy-based formula is precluded.The infant should be maintained on an elimination diet until the child is between 9-12 months of age or at least for 6 months, whichever occurs first. In most cases, symptoms will improve substantially within 2-4 weeks if diagnosis is correct. According to consensus in literature, a therapeutic formula is a formula tolerated by at least 90% (with 95% confidence) of cow's milk protein allergy infants. The primary study outcome will be the evaluation of the hypoallergenicity of a new aminoacid based formula in children with confirmed immunoglobulin (Ig)E- mediated CMA. According to the American Academy of Pediatrics (AAP) Subcommittee on Nutrition and Allergic Diseases a hypoallergenic formula must be tested in infants and children with hypersensitivity to cow's milk proteins, with findings verified by elimination-challenge tests under double-blind, placebo-controlled conditions (DBPCFC).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 1-36 months with diagnosis of Immunoglobulin E-mediated cow milk allergy in the last 12 weeks,
* full and stable remission of allergy symptoms
* Written informed consent form collected by the parents.

Exclusion Criteria:

* Infant aged <1 months and >36 months,
* breast fed infants,
* other food allergies,
* other allergic diseases,
* evidence of non-IgE-mediated CMA,
* history of severe anaphylactic reaction,
* eosinophilic disorders of the gastrointestinal tract,
* chronic systemic diseases,
* congenital cardiac defects,
* active tuberculosis,
* autoimmune diseases,
* immunodeficiency,
* chronic inflammatory bowel diseases,
* celiac disease,
* cystic fibrosis,
* metabolic diseases,
* malignancy,
* chronic pulmonary diseases,
* malformations of the gastrointestinal and/or respiratory tract,
* use of systemic antibiotics or anti-mycotic drugs during 4 weeks before study entry;
* investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements;
* participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.

Ages: 1 Month to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects tolerants to a new hypoallergenic formula demonstrated by oral food challenge with the new study formula | After one week from the oral food challenge
  All subjects perform an oral food challenge with the new study formula. If the infant not react to the new hypoallergenic formula during the oral food challenge, the subjects tolerate this product.

SECONDARY OUTCOMES:
Evaluation of body weight in children assuming amino acid based formula | after 180 days
  In the absence of reaction to the new amino acid based formula, a subgroup of child (n=15) will continue the second part of the study, with an open-label feeding with amino acid based formula for 180 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Rita Nocerino, Portici, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nocerino R, Di Scala C, Coppola S, Giglio V, Carucci L, Cosenza L, Voto L, Iannicelli AM, Luzzetti A, Berni Canani R. Tolerability of a new amino acid-based formula for children with IgE-mediated cow's milk allergy. Ital J Pediatr. 2021 Jul 3;47(1):151. doi: 10.1186/s13052-021-01096-3. PMID 34217356